CLINICAL TRIAL: NCT00632593
Title: Prospective Randomized Trial Comparing Early Complications of Hand-Sewn Versus Circular Stapled Gastro-Jejunal Anastomosis in Laparoscopic Gastric Bypass
Brief Title: Trial Comparing Early Complications of Two Techniques in the Laparoscopic Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Leonardo J Silvio, University Hospital of Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BPGlap1
Record Dates: First submitted 2008-02-28; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Obesity
Keywords: Early Complications of both techniques; Fistula rate; Dehiscence rate; reoperation rate and cause
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Circular Stapled (Active Comparator): Patients operated performing the gastric pouch of the gastric bypass with a circular staple device
  Interventions: Procedure: Laparoscopic Gastric Bypass
- Handsewn anastomosis (Active Comparator): Patients operated performing the gastric pouch of the gastric bypass in a handsewn manner
  Interventions: Procedure: Laparoscopic Gastric Bypass

INTERVENTIONS:
Procedure: Laparoscopic Gastric Bypass
  Arms: Circular Stapled
Procedure: Laparoscopic Gastric Bypass
  Arms: Handsewn anastomosis

SUMMARY:
The purpose of this study is to define and evaluate the early complications between two different surgical techniques used to perform a laparoscopic gastric bypass

ELIGIBILITY:
Inclusion Criteria:

* Body mass Index between 35 with comorbidities and 50 kg/mt2

Exclusion Criteria:

* Body mass index <35kg7mt2 and >50kg/mt2

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo J Silvio, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- University Hospital Of Bellvitge, Barcelona, Catalonia, Spain